CLINICAL TRIAL: NCT01141153
Title: Test of Efficacy and Safety of the Dual Antiplatelet Therapy Compared to the Combination of Oral Anticoagulant Therapy + Dual Antiplatelet Therapy in Patients With Atrial Fibrillation With Low-moderate Risk Submitted to Coronary Stent Implantation
Brief Title: Anticoagulation in Stent Intervention
Acronym: MUSICA-2
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MUSICA-2; 2009-017256-27 (EudraCT Number)
Record Dates: First submitted 2010-06-09; First posted 2010-06-10 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-02

CONDITIONS: Atrial Fibrillation; Stroke
Keywords: atrial fibrillation; Coronary Stent implantation; Low-moderate risk of stroke; dual antiplatelet therapy; anticoagulation
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — Aspirin; Clopidogrel; Acenocoumarol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral anticoagulation plus dual antiplatelet therapy (Experimental)
  Interventions: Drug: Acetylsalicylic Acid + clopidogrel + acenocoumarol
- Dual antiplatelet therapy (Active Comparator)
  Interventions: Drug: Acetylsalicylic Acid + clopidogrel

INTERVENTIONS:
Drug: Acetylsalicylic Acid + clopidogrel + acenocoumarol — Acetylsalicylic Acid 100 mg daily + Clopidogrel 75 mg daily + Acenocoumarol dosage with INR monitoring
  Treatment : 6 weeks for bare metal stent and 12 months for drug elution stent
  Arms: Oral anticoagulation plus dual antiplatelet therapy
Drug: Acetylsalicylic Acid + clopidogrel — Salicylic Acid, 300 mg daily + Clopidogrel 75 mg daily
  Treatment : 6 weeks for bare metal stent and 12 months for drug elution stent.
  Arms: Dual antiplatelet therapy

SUMMARY:
Objective:

The main objective is to evaluate the pattern of dual antiplatelet therapy (aspirin, 300 mg / day + clopidogrel 75 mg / day) compared to the use of the triple regimen (Acenocoumarol as control + acetylsalicylic acid 100 mg / day + Clopidogrel 75 mg / day) in patients with atrial fibrillation, low-moderate risk of stroke (CHADS ≤ 2) who are undergoing PCI-S.

Design:

Randomized, parallel, with two arms, blind evaluation by third parties.

Patients:

304 patients undergoing PCI-S with atrial fibrillation, low-moderate risk of stroke (CHADS ≤ 2), which requires prevention of thrombosis

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes older than 18 years.
* Patients with permanent atrial fibrillation, persistent or paroxysmal (at least one episode), documented electrocardiographically and receiving oral anticoagulation. Patients with acute coronary syndrome or stable angina who are undergoing PCI-S.
* Patients who have previously given their informed consent to participation in the study.

Exclusion Criteria:

* Patients who can not be followed by the research team during the 12 months provided for monitoring.
* Patients with renal failure or serum creatinine above 2 mg • dL-1, neurological deficits, active ulcer or epigastric pain.
* Patients who continue regular treatment with NSAIDs or other analgesics or corticosteroids.
* Patients undergoing reoperation.
* Patients who during the study period, should receive, according to medical criteria, other adjuvant drug treatment than that specified in this protocol.
* Pregnant women.
* Use of investigational agents or not registered within 30 days of entry into the study.
* Patients with a history of allergy to study drugs or excipients.
* Patients with severe valve disease.
* Patients with CHADS> 2.
* Patients who can not use the study drug orally.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2010-06; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
A composite of stroke, myocardial infarction, systemic thromboembolism, stent thrombosis and death | until 12 months
  Incidence of the composite major events (stroke, myocardial infarction, systemic thromboembolism, stent thrombosis and death) until 12 months after the initial treatment

SECONDARY OUTCOMES:
Incidence of major and minor bleeding | until 12 months
Adverse events | until 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Antonia Sambola, MD Ph, Principal Investigator; David García -Dorado, MD Ph, Study Director
Locations (11):
- Spain (11):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Sant Pau, Barcelona, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Corporación Sanitaria Parc Taulí, Sabadell, Barcelona
  - Hospital Marqués de Valdecilla, Santander, Cantabria
  - Hospital Dr.Josep Trueta, Girona, Girona
  - Hospital Universitario Gregorio Marañón, Madrid, Madrid
  - Hospital San Carlos, Madrid, Madrid
  - Hospital Puerta del Hierro, Majadahonda, Madrid
  - Hospital Clínic de Barcelona, Barcelona

REFERENCES:
- [Derived] Sambola A, Montoro JB, Del Blanco BG, Llavero N, Barrabes JA, Alfonso F, Bueno H, Cequier A, Serra A, Zueco J, Sabate M, Rodriguez-Leor O, Garcia-Dorado D. Dual antiplatelet therapy versus oral anticoagulation plus dual antiplatelet therapy in patients with atrial fibrillation and low-to-moderate thromboembolic risk undergoing coronary stenting: design of the MUSICA-2 randomized trial. Am Heart J. 2013 Oct;166(4):669-75. doi: 10.1016/j.ahj.2013.07.028. Epub 2013 Sep 14. PMID 24093846